CLINICAL TRIAL: NCT03395964
Title: Comparison of Preoperative CT Scan Guided and Intraoperative Hybrid DynaCT Scan-Guided Small Lung Tumor Localization: A Randomized Study
Brief Title: Comparison of Preoperative CT Scan Guided and Intraoperative Hybrid DynaCT Scan-Guided Small Lung Tumor Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-IRB-201600671A3
Record Dates: First submitted 2017-11-29; First posted 2018-01-10 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-01

CONDITIONS: Small and/or Deep Lung Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative CT scan-guided localization (Active Comparator): Preoperative localization of the lung nodule will be carried out in the radiology department on the day of surgery using local anesthesia. CT-guided hook-wire or methyl blue dye will be placed percutaneously through a 22-gauge needle with the distal end deep to the nodule. The patient will then be taken to the operating room, where under general anesthesia with lung isolation, the nodule will be removed by wedge excision with endostaplers (Endo-GIA-II, United States Surgical,Norwalk, Conn; Echelon Endostapler, Ethicon Endo-Surgery, Cincinnati,Ohio) under the guidance of preoperative lung marking. If the lesion could not be excised using the VATS technique, the patient underwent an open thoracotomy.
  Interventions: Procedure: Preoperative CT scan-guided localization
- Hybrid Dyna-CT guided localization (Experimental): Patients will be brought into the Hybrid OR, and placed in the lateral decubitus position. A C-arm CT scan of the pre-determined ﬁeld of view that included the nodule position will be acquired during an end-inspiratory hold maneuver using a 5 sec scan protocol with 0.36mGy/projection and 248 projections acquired over 200°. The radiologist reviewed the C-arm CT scan to localize the nodule and plan trajectories for percutaneous hook-wire placement using Syngo iGuide needle guidance software. The planned needle pathways will be integrated into the C-arm fluoroscopic imaging system, which provided laser crossbar and guidance markers on fluoroscopy images to direct the needle pathway for hook wire placement.
  Interventions: Procedure: Hybrid Dyna-CT guided localization

INTERVENTIONS:
Procedure: Hybrid Dyna-CT guided localization — We will perform intraoperative lung tumor localization in CGMH hybrid operation room(Room 51) equipped with the Siemens Artis Zeego system with DynaCT imaging capabilities. The system provides images equivalent to a 16-slice spiral CT scanner in a single 6-s sweep.
  Arms: Hybrid Dyna-CT guided localization
Procedure: Preoperative CT scan-guided localization — Preoperative localization of the lung nodule will be carried out in the radiology department on the day of surgery using local anesthesia. CT-guided hook-wire or methyl blue dye will be placed percutaneously through a 22-gauge needle with the distal end deep to the nodule. The patient will then be taken to the operating room, where under general anesthesia with lung isolation, the nodule will be removed by wedge excision with endostaplers (Endo-GIA-II, United States Surgical,Norwalk, Conn; Echelon Endostapler, Ethicon Endo-Surgery, Cincinnati,Ohio) under the guidance of preoperative lung marking. If the lesion could not be excised using the VATS technique, the patient underwent an open thoracotomy.
  Arms: Preoperative CT scan-guided localization

SUMMARY:
It is well known that video-assisted thoracoscopic surgery(VATS) is preferred to open surgery for lung resection because of the use of smaller incisions and optimized postoperative recovery, including a shorter length of hospitalization. Studies have shown decreased operative and post-operative morbidity with decreased operative times. However, for small nodules (i.e. lesions <1 cm or those at a distance more than 1.5cm from the lung periphery), adequate identification of the target nodule has been be difficult by VATS, and a more significant resection or conversion to thoracotomy is occasionally needed to ensure complete resection.

In order to improve nodule localization, a variety of preoperative localization methods such as CT-guide hook wire or methyl blue dye localization have been proposed and described to mark lung nodules for easier identification of small nodules and help guide resection during VATS. However, there are certain concerns. First, there are the difficult logistics in minimizing the time between the localization procedure and the subsequent surgery. Second, there is concern for patient safety, in particular pneumothorax, during transfer to and from the ward to the radiology department and in the frequent delays and waiting in reception areas prior to transfer to operating heaters. Finally, interdepartmental transfers and delays can also increase the risk of hook-wire dislodgement.

Theoretically, the aforementioned disadvantage could be solved by performing the localization procedure and the lung surgery in the same hybrid operating room environment.

In the current study, the investigators will perform intraoperative lung tumor localization in CGMH hybrid operation room (Room 51) equipped with the Siemens Artis Zeego system with DynaCT imaging capabilities. The system provides images equivalent to a 16-slice spiral CT scanner in a single 6-s sweep. Through a randomized study design, the advantages, disadvantages, and important considerations of this combined approach will be compared with traditional preoperative CT scan guided localization protocol.

DETAILED DESCRIPTION:
Lung Cancer continues to have high morbidity and mortality, and it is estimated that in 2014 in Taiwan there were approximately 11692 new cases and 9167 deaths from lung cancer, which was the first leading cause of cancer deaths. Because 70% of lung cancer patients in Taiwan were diagnosed at late stage, only palliative treatment could be given and prognosis was poor.

Owing so, screening and early detection of early stage lung cancer is of paramount importance. In 2012, the National Lung Screening Trial demonstrated that screening for lung cancer with chest computed tomography (CT) results in a 20% reduction in mortality. Low dose CT(LDCT) has been acknowledged as the most powerful tool for early lung cancer detection. With the increasing use of CT, it is expected that many patients with small lesions (< 2 cm), enlarging lesions, and partially solid lesions that are suspicious for cancer will be discovered and will require surgical resection.

It is well known that video-assisted thoracoscopic surgery(VATS) is preferred to open surgery for lung tumor resection because of the use of smaller incisions and optimized postoperative recovery, including a shorter length of hospitalization. Studies have shown decreased operative and post-operative morbidity with decreased operative times. While this procedure speeds up recovery and potentially reduces complications, the loss of natural vision and tactile sensing makes it difficult for the surgeon to locate the nodules, especially in cases of non-superficial, ground-glass opaque, and small lesions. The yield rate for nodules < 1 cm can be below 40% as studies show. And a more significant resection (more healthy tissue is resected than actually necessary in order to avoid missing the lesion.) or conversion to thoracotomy is occasionally needed to ensure complete resection. In order to improve nodule localization, a variety of methods have been proposed and described to mark lung nodules for easier identification of small nodules and help guide resection during VATS. These ranged from percutaneous image guided injection of a dye (methylene blue) or radio-opaque material such as barium sulphate, to percutaneously placed hookwires and micro-coils in the radiology suite prior to surgery. All these preoperative CT scan guided localization procedures were carried out "outside" operation room and under local anesthesia.

However, there remain certain concerns. First, there are the difficult logistics in minimizing the time between the hookwire procedure and the subsequent surgery. Second, there is concern for patient safety, in particular pneumothorax, during transfer to and from the ward to the radiology department and in the frequent delays and waiting in reception areas prior to transfer to operating theaters. Finally, interdepartmental transfers and delays can also increase the risk of hookwire dislodgement.

Theoretically, the aforementioned disadvantage could be solved by performing the localization procedure and the lung surgery in the same hybrid operating room environment(i.e. Hybrid OR). A hybrid operating room is a surgical theatre that is equipped with advanced medical imaging devices such as fixed C-Arms, CT scanners or MRI scanners. These imaging devices enable minimally-invasive surgery, which is less traumatic for the patient.

Hybrid operating rooms are currently used mainly in cardiac, vascular and neuro-surgery, and could be suitable for a number of other surgical disciplines, such as thoracic surgery.

Using advanced intra-operative imaging in the OR helps to precisely locate and resect the lesion in a potentially tissue-sparing and quick fashion. In order to be able to use image guidance during VATS, rotational angiography has to be performed before the introduction of ports, thus before the lobe in question deflates. This way the lesion is visible through the natural contrast of air. In a second step, hook wires, thread needles, or contrast agent (Lipiodol, Iopamidol) are introduced into or next to the lesion to ensure visibility on the angiogram after lung deflation. Then, the conventional part of VATS starts with the introduction of thoracoscope. The imaging system is used in fluoroscopic mode now, where both the inserted instruments and the previously marked lesion are well visible. A precise resection is now possible. In case contrast agent has been used to mark the lesion, it will also drain into the regional lymph nodes, which then can be resected within the same procedure.

Reviewing the literature, there are several studies reporting the efficacy of Hybrid OR in localization of the lung nodule with good result and acceptable radiation exposure. However, there was no study so far comparing the efficacy of intraoperative localization and preoperative CT guided localization.

In the current study, the investigators will perform intraoperative lung tumor localization in CGMH hybrid OR(Room 51) equipped with the Siemens Artis Zeego system with DynaCT imaging capabilities. The system provides images equivalent to a 16-slice spiral CT scanner in a single 6-s sweep. Through a randomized study design, the advantages, disadvantages, and important considerations of this combined approach will be compared with traditional preoperative CT scan guided localization protocol.

ELIGIBILITY:
Inclusion Criteria:

* lesions <1 cm or those at a distance more than 1.5cm from the lung periphery.

Exclusion Criteria:

* confirmed as a malignancy
* Age <18
* serious pulmonary heart disease
* more than one tumors needed localization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Procedure time | from initiation of the preprocedural CT scanning to the end of the postprocedural CT scanning, through study completion, an average of 2 year.
  Recording the time of localization procedure, including needle puncture time.

SECONDARY OUTCOMES:
Complications | Beginning from localization until operation, through study completion, an average of 2 year.
  pneumothorax and hemorrhage
Radiation dose | from initiation of the preprocedural CT scanning to the end of the postprocedural CT scanning, through study completion, an average of 2 year.
  Effective dose estimates were performed using thermoluminescent dosimeters (TLD).

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Kai Chao, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang BY, Huang JY, Cheng CY, Lin CH, Ko J, Liaw YP. Lung cancer and prognosis in taiwan: a population-based cancer registry. J Thorac Oncol. 2013 Sep;8(9):1128-35. doi: 10.1097/JTO.0b013e31829ceba4. PMID 23945383
- [Background] Huang HL, Kung PT, Chiu CF, Wang YH, Tsai WC. Factors associated with lung cancer patients refusing treatment and their survival: a national cohort study under a universal health insurance in Taiwan. PLoS One. 2014 Jul 7;9(7):e101731. doi: 10.1371/journal.pone.0101731. eCollection 2014. PMID 24999633
- [Background] Bach PB, Mirkin JN, Oliver TK, Azzoli CG, Berry DA, Brawley OW, Byers T, Colditz GA, Gould MK, Jett JR, Sabichi AL, Smith-Bindman R, Wood DE, Qaseem A, Detterbeck FC. Benefits and harms of CT screening for lung cancer: a systematic review. JAMA. 2012 Jun 13;307(22):2418-29. doi: 10.1001/jama.2012.5521. PMID 22610500
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] National Lung Screening Trial Research Team; Church TR, Black WC, Aberle DR, Berg CD, Clingan KL, Duan F, Fagerstrom RM, Gareen IF, Gierada DS, Jones GC, Mahon I, Marcus PM, Sicks JD, Jain A, Baum S. Results of initial low-dose computed tomographic screening for lung cancer. N Engl J Med. 2013 May 23;368(21):1980-91. doi: 10.1056/NEJMoa1209120. PMID 23697514
- [Background] Oken MM, Hocking WG, Kvale PA, Andriole GL, Buys SS, Church TR, Crawford ED, Fouad MN, Isaacs C, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Ragard LR, Rathmell JM, Riley TL, Wright P, Caparaso N, Hu P, Izmirlian G, Pinsky PF, Prorok PC, Kramer BS, Miller AB, Gohagan JK, Berg CD; PLCO Project Team. Screening by chest radiograph and lung cancer mortality: the Prostate, Lung, Colorectal, and Ovarian (PLCO) randomized trial. JAMA. 2011 Nov 2;306(17):1865-73. doi: 10.1001/jama.2011.1591. Epub 2011 Oct 26. PMID 22031728
- [Background] Humphrey LL, Deffebach M, Pappas M, Baumann C, Artis K, Mitchell JP, Zakher B, Fu R, Slatore CG. Screening for lung cancer with low-dose computed tomography: a systematic review to update the US Preventive services task force recommendation. Ann Intern Med. 2013 Sep 17;159(6):411-420. doi: 10.7326/0003-4819-159-6-201309170-00690. PMID 23897166
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for lung cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 4;160(5):330-8. doi: 10.7326/M13-2771. PMID 24378917
- [Background] Suzuki K, Nagai K, Yoshida J, Ohmatsu H, Takahashi K, Nishimura M, Nishiwaki Y. Video-assisted thoracoscopic surgery for small indeterminate pulmonary nodules: indications for preoperative marking. Chest. 1999 Feb;115(2):563-8. doi: 10.1378/chest.115.2.563. PMID 10027460
- [Background] Santambrogio R, Montorsi M, Bianchi P, Mantovani A, Ghelma F, Mezzetti M. Intraoperative ultrasound during thoracoscopic procedures for solitary pulmonary nodules. Ann Thorac Surg. 1999 Jul;68(1):218-22. doi: 10.1016/s0003-4975(99)00459-2. PMID 10421144
- [Background] Kim YD, Jeong YJ, I H, Cho JS, Lee JW, Kim HJ, Lee SH, Kim DH. Localization of pulmonary nodules with lipiodol prior to thoracoscopic surgery. Acta Radiol. 2011 Feb 1;52(1):64-9. doi: 10.1258/ar.2010.100307. PMID 21498328
- [Background] Mayo JR, Clifton JC, Powell TI, English JC, Evans KG, Yee J, McWilliams AM, Lam SC, Finley RJ. Lung nodules: CT-guided placement of microcoils to direct video-assisted thoracoscopic surgical resection. Radiology. 2009 Feb;250(2):576-85. doi: 10.1148/radiol.2502080442. PMID 19188326
- [Background] Finley RJ, Mayo JR, Grant K, Clifton JC, English J, Leo J, Lam S. Preoperative computed tomography-guided microcoil localization of small peripheral pulmonary nodules: a prospective randomized controlled trial. J Thorac Cardiovasc Surg. 2015 Jan;149(1):26-31. doi: 10.1016/j.jtcvs.2014.08.055. Epub 2014 Sep 16. PMID 25293355
- [Background] Kpodonu J, Raney A. The cardiovascular hybrid room a key component for hybrid interventions and image guided surgery in the emerging specialty of cardiovascular hybrid surgery. Interact Cardiovasc Thorac Surg. 2009 Oct;9(4):688-92. doi: 10.1510/icvts.2009.209429. Epub 2009 Jul 21. PMID 19622541
- [Background] Biasi L, Ali T, Ratnam LA, Morgan R, Loftus I, Thompson M. Intra-operative DynaCT improves technical success of endovascular repair of abdominal aortic aneurysms. J Vasc Surg. 2009 Feb;49(2):288-95. doi: 10.1016/j.jvs.2008.09.013. Epub 2008 Nov 28. PMID 19038527
- [Background] Heran NS, Song JK, Namba K, Smith W, Niimi Y, Berenstein A. The utility of DynaCT in neuroendovascular procedures. AJNR Am J Neuroradiol. 2006 Feb;27(2):330-2. PMID 16484404
- [Background] Irie K, Murayama Y, Saguchi T, Ishibashi T, Ebara M, Takao H, Abe T. Dynact soft-tissue visualization using an angiographic C-arm system: initial clinical experience in the operating room. Neurosurgery. 2008 Mar;62(3 Suppl 1):266-72; discussion 272. doi: 10.1227/01.neu.0000317403.23713.92. PMID 18424996
- [Background] Gill RR, Zheng Y, Barlow JS, Jayender J, Girard EE, Hartigan PM, Chirieac LR, Belle-King CJ, Murray K, Sears C, Wee JO, Jaklitsch MT, Colson YL, Bueno R. Image-guided video assisted thoracoscopic surgery (iVATS) - phase I-II clinical trial. J Surg Oncol. 2015 Jul;112(1):18-25. doi: 10.1002/jso.23941. Epub 2015 May 28. PMID 26031893
- [Background] Ng CSH, Man Chu C, Kwok MWT, Yim APC, Wong RHL. Hybrid DynaCT scan-guided localization single-port lobectomy. [corrected]. Chest. 2015 Mar;147(3):e76-e78. doi: 10.1378/chest.14-1503. PMID 25732474
- [Background] Rouze S, de Latour B, Flecher E, Guihaire J, Castro M, Corre R, Haigron P, Verhoye JP. Small pulmonary nodule localization with cone beam computed tomography during video-assisted thoracic surgery: a feasibility study. Interact Cardiovasc Thorac Surg. 2016 Jun;22(6):705-11. doi: 10.1093/icvts/ivw029. Epub 2016 Feb 26. PMID 26921886
- [Derived] Chao YK, Pan KT, Wen CT, Fang HY, Hsieh MJ. Preoperative CT versus intraoperative hybrid DynaCT imaging for localization of small pulmonary nodules: a randomized controlled trial. Trials. 2019 Jul 4;20(1):400. doi: 10.1186/s13063-019-3532-z. PMID 31272483